CLINICAL TRIAL: NCT06758531
Title: Coffee Bioequivalence Trial: Comparing the Pharmacokinetics of Bioactive Components and Physiological Effects of Consuming Encapsulated Instant Coffee Versus Traditional Instant Coffee Brewed in Water
Brief Title: Coffee Bioequivalence Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Charlotte E Mills, Hugh Sinclair Lecturer in Nutritional Sciences, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 24/28
Record Dates: First submitted 2024-11-18; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Liver Functions; Bioequivalence; Cardiovascular Risk; Cardiometabolic Risk Markers
Keywords: Coffee; Bioequivalence; Caffeine; Liver function; Polyphenols; Blood pressure; Cardiovascular disease; Chlorogenic acids
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Coffee given as a drink (Active Comparator): This group will consume 3.6 g of commercially available instant coffee given as a drink prepared with 400 ml of water.
  Interventions: Dietary Supplement: Instant coffee given as a drink
- Coffee given in tablet form (Active Comparator): This group will receive 3.6 g of instant coffee provided as 4 tablets consumed with 400 ml of water.
  Interventions: Dietary Supplement: Coffee given in a tablet form
- Control group (Placebo Comparator): The caffeine free coffee control will be provided as 4 tablets given with 400 ml of water.
  Interventions: Dietary Supplement: Control (placebo)

INTERVENTIONS:
Dietary Supplement: Instant coffee given as a drink — Commercially available instant coffee (3.6 g) will be provided in the form of a drink prepared with 400 ml of water. A standard breakfast consisting of cereal with milk will be provided at 60 mins after the intervention. A standard lunch (cheese sandwiches, potato crisps and shortbread biscuits) will be given at 300 after coffee intake.
  Arms: Coffee given as a drink
Dietary Supplement: Coffee given in a tablet form — Commercially available instant coffee (3.6 g) will be provided as 4 tablets given with 400 ml of water. A standard breakfast consisting of cereal with milk will be provided at 60 mins after the intervention. A standard lunch (cheese sandwiches, potato crisps and shortbread biscuits) will be given at 300 after coffee intake.
  Arms: Coffee given in tablet form
Dietary Supplement: Control (placebo) — A caffeine and coffee free control (3.6 g) will be provided as 4 tablets given with 400 ml of water. A standard breakfast consisting of cereal with milk will be provided at 60 mins after the intervention. A standard lunch (cheese sandwiches, potato crisps and shortbread biscuits) will be given at 300 after coffee intake.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to test if coffee consumed as a tablet is biologically equivalent to that consumed traditionally as a drink. It will also learn about the impact of the short-term intake of coffee on markers of cardiovascular and liver health. The main questions it aims to answer are:

* Do coffee bioactive compounds produce the same levels in blood and urine regardless of how the coffee is consumed (tablet or drink)?
* How does coffee as a tablet or drink impact cardiovascular risk and liver health versus a non-coffee control?

Participants will:

* Visit the clinical unit for three phases; each phase is 1x 480 minute (eight hour) acute postprandial visit and 1 x one hour visit the following day. During each phase they will be randomly assigned to take a different intervention (coffee drink, coffee tablet, coffee-free control)
* Be cannulated during the 480 minute (8 hour) acute visits and have regular blood draws as well as basic clinical assessments
* Return on day two for a fasting blood sample and basic clinical assessment
* Collect their urine for 24 h
* Be asked to record their intake of foods and drinks for 3 days to assess their usual diet (dietary assessment).

DETAILED DESCRIPTION:
Coffee has gained interest for its role in the prevention of non-communicable diseases such as heart and liver diseases. Population-based studies have reported that consuming 2-4 cups of coffee per day is associated with lower death rates and, notably reductions in the incidence of heart disease. However, these observational trials do not directly prove causality and carefully designed randomised controlled trials are needed.

This current trial will provide vital information to inform a large-scale randomised controlled trial assessing the effects of coffee consumption on risk markers for developing cardiometabolic disease (such as type 2 diabetes, heart and liver diseases) to test causality. In this follow-up trial to be conducted in 2025, non-coffee consumers will be recruited. To maximise recruitment, retention and adherence in the trial, we are considering providing instant coffee as tablets rather than as a drink. Hence, the current study will help to understand if coffee delivered in a tablet is biologically equivalent to consuming coffee as a drink.

A 3 armed, randomised, controlled crossover trial in healthy participants wil be performed. The primary outcome is the pharmacokinetic profile of coffee bioactives in coffee drink versus the coffee tablet. Secondary outcomes will be assessing the impact of the coffee both as a drink and tablet on cardiovascular and liver health markers (versus a coffee-free control).

Briefly, participants will attend three study phases. Each study phase includes a 480 minute (8-hour) acute postprandial visit and a shorter visit (~one hour) the following morning. On the first day participants will arrive having fasted overnight and having followed dietary and lifestyle restrictions in the preceding days. They will have baseline anthropometric measures performed and a cannula will be inserted; two baseline blood samples will be collected (14 mL in total). Blood samples will be collected regularly from the cannula, and a clinic blood pressure measurement will be performed at regular intervals following the intervention (a different intervention will be given in a random order at each of the three phases). A breakfast meal and lunch will be provided to the participants during the visit and participants will leave with a standardised meal and snack to consume in the evening. They will return, fasted the following morning to provide a blood samples and have their blood pressure measured. Participants will be asked to collect their urine for 24h following the intervention; this will be returned that morning. There will be a 4-week period between each study phase.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and pre-menopausal females (must have regular menstrual cycles)
* Aged between 18 to 45 years
* Body mass index (BMI) between 18.5-30 kg/m2

Exclusion Criteria:

* Sensitivity to coffee and caffeine
* Food allergies relating to the test meals provided (such as gluten or lactose intolerance)
* Current smoking and vaping use.
* Medical history of chronic diseases (cancer, high blood pressure (hypertension), type 2 diabetes, heart attack and/or any other heart disease related diseases, gastrointestinal disorders, hyperlipidaemia, kidney or liver disease).
* Diagnosed with anaemia
* Prescribed any medication relating to the study outcome measures (such as blood pressure lowering, anti-inflammatories or blood thinners).
* Drinking more than the recommended intake for alcohol (> 14 units/week)
* Taking any supplements (vitamins, minerals, probiotics).
* Any other unusual medical history or diet and lifestyle habits or practices that would preclude volunteers from participating in a dietary intervention and metabolic study (e.g. pacemaker)
* Planning on a weight-reducing regimen (lost >3 kg in the last 6 months)
* Parallel participation in another intervention study
* Pregnancy, planning a pregnancy in the next 6 months or breastfeeding
* NHS blood donation in the last 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic profile of key coffee biologically active compounds and their metabolites after consuming a coffee drink, a coffee tablet and control. | Blood taken prior to consuming the intervention (0 minutes) and then 30, 45, 60, 90, 120, 180, 240, 300, 360, 420, 480 and 1440 minutes post intervention.
  Key coffee biologically active compounds and their metabolites (e.g. chlorogenic acids, caffeine, trigonelline) will be measured in plasma samples collected over a 24 h period after each intervention. The pharmacokinetic profile (absorption, metabolism and excretion), maximal concentration, Cmax will be calculated.
Pharmacokinetic profile of key coffee biologically active compounds and their metabolites after consuming a coffee drink, a coffee tablet and control. | Blood taken prior to consuming the intervention (0 minutes) and then 30, 45, 60, 90, 120, 180, 240, 300, 360, 420, 480 and 1440 minutes post intervention.
  Key coffee biologically active compounds and their metabolites (e.g. chlorogenic acids, caffeine, trigonelline) will be measured in plasma samples collected over a 24 h period after each intervention. The pharmacokinetic profile (absorption, metabolism and excretion), area under the concentration curve will be calculated.

SECONDARY OUTCOMES:
Fasting concentrations of total cholesterol and high-density lipoprotein cholesterol. | Acute study days prior to the intervention (0 minutes).
  Serum lipids will be measured directly using a clinical chemistry analyser.
Fasting and postprandial lipids concentrations after consuming the coffee drink, coffee tablet and control interventions | Acute study days, blood taken prior to the intervention (0 minutes) and then 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 420 and 480 minutes.
  Serum triacylglycerol and non-esterified fatty acids will be measured in the fasting and postprandial blood samples collected for 480 min after each intervention.
Fasting and postprandial glucose concentrations after consuming the coffee drink, coffee tablet and control interventions | Acute study days, blood taken prior to consuming the intervention (0 minutes) and then 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 420 and 480 minutes.
  Serum glucose will be measured in the acute study day blood samples collected for 480 minutes after each intervention using a clinical chemistry analyser.
Fasting and postprandial insulin concentrations after consuming the coffee drink, coffee tablet and control interventions | Acute study days, blood taken prior to consuming the intervention (0 minutes) and then 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 420 and 480 minutes.
  Serum insulin will be measured in the acute study day blood samples collected for 480 minutes after each intervention using an enzyme-lined immunosorbent assay.
Fasting and postprandial liver enzyme concentrations after consuming the coffee drink, coffee tablet and control interventions | Acute study days, blood taken prior to consuming the intervention (0 minutes) and then 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 420 and 480 minutes.
  Serum alanine transaminase (ALT), aspartate transferase (AST), alkaline phosphatase (ALP), gamma-glutamyl transferase (GGT) and glutamate dehydrogenase (GLDH) will be measured in the acute study day blood samples collected for 480 minutes after each intervention using a clinical chemistry analyser.
Fasting and postprandial gut hormone concentrations after consuming the coffee drink, coffee tablet and control interventions | Acute study days, blood taken prior to the intervention (0 minutes) and then 30, 60, 120, 180, 240, 300, 360 and 480 minutes.
  C-peptide, GIP, GLP-1 and Ghrelin will be measured in the postprandial blood samples collected for 480 min after each interventions.
Fasting and postprandial plasma metabolomics after consuming the coffee drink, coffee tablet and control interventions | Acute study days, blood taken prior to the intervention (0 minutes) and then 30, 60, 120, 180, 240, 300, 360, 420 and 480 minutes.
  Metabolomics will be measured in the postprandial blood samples collected for 480 min after the interventions using NMR.
Fasting and postprandial plasma nitrate and nitrite concentrations after consuming the coffee drink, coffee tablet and control interventions | Acute study days, blood taken prior to the intervention (0 minutes) and then 15, 30, 45, 60, 120, 180, 240, 300, 360, 420 and 480 minutes.
  Nitrate, nitrite and Nox (sum of nitrate and nitrite) will be measured in the postprandial blood samples collected for 480 min after each intervention.
Urinary metabolomics | Urine will be collected prior to (0 minutes) and for 1440 minutes after each intervention.
  Metabolomics will be performed on the 24 h urine samples using NMR .
Urinary creatinine | Urine will be collected prior to (0 minutes) and for 1440 minutes after each intervention.
  Creatinine will be measured in the 24 h urine samples using a clinical chemistry analyser.
Urinary osmolality and pH | Urine will be collected prior to (0 minutes) and for 1440 minutes after each intervention.
  Osmolality will be determined as a measure of the concentration of solutes in the 24 h urine sample and pH to indicate whether the sample is acidic or alkaline after consuming the study interventions.
Urinary sodium and potassium | Urine will be collected prior to (0 minutes) and for 1440 minutes after each intervention.
  Sodium and potassium will be determined in the 24 h urine sample as a marker of kidney function and a nutritional biomarker after consuming the study interventions.
Body weight | On each acute study visit prior to the collection of the first blood sample (0 minutes).
  Body weight will be measured using a Tanita scale.
Height | First acute study visit (0 minutes on visit 1)
  Height will be measured to the nearest cm using a stadiometer
Blood pressure | -15, 30, 60, 120, 180, 240, 300, 360, 420, 480 minutes
  Blood pressure will be measured using blood pressure monitor.
Body fat percentage | Each acute study visit (0 minutes)
  Body fat percentage will be measured using the Tanita scale by bioelectrical impedance.
Body fat mass | On each acute study visit prior to the collection of the first blood sample (0 minutes).
  Body fat mass will be measured using a Tanita scale.
Body lean mass | On each acute study visit prior to the collection of the first blood sample (0 minutes).
  Body lean mass will be measured using a Tanita scale.
Body mass index | On each acute study visit (0 minutes)
  Body mass index will be calculated using the body weight (kg) and height (m) data.
Waist and hip circumferences | On each acute study visit (0 minutes).
  A non-stretch tape will be used to measure waist and hip circumferences
Habitual dietary intake of the study participants | Two weeks prior to the first acute study visit (t- 2 weeks from visit 1).
  Record of the food and drink prior to the first study visit
Fasting estimate of insulin resistance and insulin sensitivity | On each acute study visit (0 minutes).
  HOMA-IR (Homeostasis model assessment estimated insulin resistance) and QUICKI (Quantitative Insulin Sensitivity Check Index) will be calculated using the fasting glucose and insulin data.
Fasting low-density lipoprotein-cholesterol concentration | On each acute study visit (0 minutes).
  The low-density lipoprotein-cholesterol concentration will be calculated from aforementioned outcomes using the Friedewald formula.

CONTACTS AND LOCATIONS:
Overall Officials: Abbe Davy, BSc, Study Director — University of Reading
Locations (1):
- Hugh Sinclair Unit of Human Nutrition, Department of Food and Nutritional Sciences, University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All anonymised IPD that underlie the results in a publication and analytical code for the statistical analysis
Supporting Information: Study Protocol, Analytic Code
Time Frame: Anonymised data will be made available on reasonable request to the study Chief Investigator one year after manuscripts have been published.
Access Criteria: For data sharing and preservation, anonymised IPD will be archived in the University of Reading Research Data Archive. Access will be overseen by the project Chief Investigator (Dr Charlotte Mills).